CLINICAL TRIAL: NCT04974736
Title: Electronic Pediatric Office Systems to Support Treatment for Parental Tobacco Use
Brief Title: eCEASE to Support Treatment for Parental Tobacco Use
Acronym: eCEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Jonathan P. Winickoff, MD, MPH, Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P001892; 1R01CA245145-01 (NIH); 20-018146 (Other: The Children's Hospital of Philadelphia)
Record Dates: First submitted 2021-06-30; First posted 2021-07-23 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Tobacco Smoking; Second Hand Tobacco Smoke; Smoking Cessation
Keywords: Family tobacco screening; Tobacco cessation
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation; Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: 2-arm Randomized Control Trial with a stratified cluster randomization
Who Masked: Outcomes Assessor
Masking Description: After the intervention has been assigned at random to one practice in each of the six pairs, the intervention will be blinded at random with either the label "A" or the label "B", and the other label will be assigned to the control practice. The statisticians will be blinded as to which of "A" and "B" is the intervention until the analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iEHR + Navigator (Experimental)
  Interventions: Behavioral: iEHR + Navigator
- Usual Care Control (No Intervention): Usual care delivery in pediatric primary care offices.

INTERVENTIONS:
Behavioral: iEHR + Navigator — The iEHR + Navigator intervention consists of an iEHR part of the intervention in the pediatric primary care setting which will include routine screening of families for tobacco use and treatment delivery to parents who smoke and will be linked to the child's electronic health record.
  The enrolled parents will also be offered support from Community Health Navigators, who will work with offices to provide customized cessation support to tobacco users, ensuring access to medications and services.
  Arms: iEHR + Navigator

SUMMARY:
The proposed project aims to develop an innovative and disseminable electronic health record (iEHR)-based approach that supports optimal primary care workflows to routinely screen families for tobacco and e-cigarette use, address household smoking behavior and promote smoke-free and e-cigarette free home and car rules in a routine and effective manner in the pediatric setting. Additionally, parents enrolled in the study will be offered assistance by a community health navigator (CHN). This study aims to examine how effective the iEHR + Navigator strategy is compared to usual care control.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal guardians who smoke, are present at the visit, and whose child is seen by a child healthcare clinician in a participating practice. "Smoker" will be defined as answering "yes" to either of the screening questions: "Have you smoked a cigarette, even a puff, in the past 7 days?" and "Have you smoked any other tobacco product (cigars like black and mild, hookah), even a puff, in the past 7 days?"

Exclusion Criteria:

1. Parent/legal guardian does not speak English;
2. No telephone; and
3. Prior enrollment in the study during a previous visit.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 817 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, after the associated research findings have been published, we will make our dataset available to investigators who email their data analysis plan to the principal investigators with the approval the Institutional Review Board (IRB) of record at Children's Hospital of Philadelphia (CHOP) and Health Information Services Group (responsible for ensuring HIPPA compliance). The data will be de-identified and validated. The dataset will include a codebook that defines the variables and describes the structure of the dataset.
Time Frame: After the associated research findings have been published.
Access Criteria: Email to the principal investigators at CHOP and Massachusetts General Hospital (MGH).

REFERENCES:
- [Derived] Nabi-Burza E, Jenssen BP, Jeffers AM, Ramachandran J, Thayer JG, Hipple B, Levy DE, Grundmeier RW, Drouin O, Vangel M, Rigotti NA, Bryant-Stephens T, Nekrasova E, McKnight M, Winickoff JP, Fiks AG. Automated Tobacco Cessation Intervention for Parents in Pediatric Primary Care: A Cluster-Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2529384. doi: 10.1001/jamanetworkopen.2025.29384. PMID 40864466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cluster randomized controlled trial, conducted from July 2021 to August 2023 in Twelve Philadelphia region pediatric primary care practices within the Children's Hospital of Philadephia network. Parents who used combusted tobacco in the past seven days and attended a child's preventive healthcare visit were enrolled in the study.
Pre-assignment Details: A two-arm parallel cluster randomized trial was conducted in 12 pediatric practices at Children's Hospital of Philadelphia. Practices were eligible if ≥10% of child patients had Medicaid and ≥40 daily visits. Eligible practices were paired based on size and estimated smoking rate, with six pairs selected to ensure sufficient size and representativeness. Within each pair, practices were randomly assigned to either the intervention or control group using computer-generated allocation.
Units Other Than Participants: Practices
Groups:
- eCEASE (iEHR + Navigator): Parents in intervention practices were proactively offered eCEASE (automated delivery of Nicotine Replacement Therapy (NRT), enrollment in the quitline and SmokefreeTXT, and cessation support from a health navigator).
Period: Overall Study
Arm/Group | eCEASE (iEHR + Navigator) | Usual Care Control
Started | 408; 6 Practices | 409; 6 Practices
Completed | 367; 6 Practices | 368; 6 Practices
Not Completed | 41; 0 Practices | 41; 0 Practices

BASELINE CHARACTERISTICS:
Groups:
- eCEASE (iEHR + Navigator): iEHR + Navigator: The iEHR + Navigator intervention consists of an iEHR part of the intervention in the pediatric primary care setting which will include routine screening of families for tobacco use and treatment delivery to parents who smoke and will be linked to the child's electronic health record.
  The enrolled parents will also be offered support from Community Health Navigators, who will work with offices to provide customized cessation support to tobacco users, ensuring access to medications and services.
- Total: Total of all reporting groups
Arm/Group | eCEASE (iEHR + Navigator) | Usual Care Control | Total
Number analyzed (Participants) | 408 | 409 | 817
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 401 | 405 | 806
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (8.89) | 35.9 (8.454) | 36.17 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant chose to not share their sex.
  Participants
    number analyzed (Participants) | 407 | 409 | 816
    Female | 335 | 337 | 672
    Male | 72 | 72 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 28 | 68
  Not Hispanic or Latino | 368 | 381 | 749
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 17 | 3 | 20
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 165 | 179 | 344
  White | 173 | 204 | 377
  More than one race | 46 | 21 | 67
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — Parents were enrolled at 12 pediatric practices in eastern Pennsylvania.
  participants
    United States | 408 | 409 | 817

OUTCOME MEASURES:

1. Primary Outcome: Parental Combusted Tobacco Quit Rate at 12 Months
Description: Parental 7-day combusted tobacco quit rates, as assessed by validated surveys, biochemically confirmed at 12 months between the intervention & usual care arms
Time Frame: 12-months
Measure: Count of Participants; unit: Participants
Arm/Group | eCEASE (iEHR + Navigator) | Usual Care Control
Number analyzed (Participants) | 408 | 409
Participants | 34 | 26

2. Secondary Outcome: Rates of Parental Quit Attempts
Description: Rates of parents' self-reported quit attempts between the intervention & usual care control arms, assessed by validated surveys of parents
Time Frame: 12-months
Population: Those parents who completed the follow-up survey and reported smoking a tobacco product in the last 7 days were used in the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | eCEASE (iEHR + Navigator) | Usual Care Control
Number analyzed (Participants) | 278 | 299
Participants | 205 | 189

3. Secondary Outcome: Rates of Parental Use of Pharmacotherapy or Services
Description: Rates of parental use of pharmacotherapy and Quitlines between the intervention & usual care arms, assessed by validated surveys of parents
Time Frame: 12-months
Population: Participants who completed the 12 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | eCEASE (iEHR + Navigator) | Usual Care Control
Number analyzed (Participants) | 367 | 368
Participants
  Used Nicotine Replacement Therapy | 177 | 59
  Enrolled in quitline | 79 | 11
  Enrolled in SmokefreeTXT | 71 | 9

4. Secondary Outcome: Rates of Parental Institution of Smoking and Vaping Bans in Their Homes and Cars
Description: Rates of parental institution of smoking and vaping bans in their homes and cars between the intervention & usual care arms, assessed by validated surveys of parents
Time Frame: 12-months
Population: Participants who completed follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | eCEASE (iEHR + Navigator) | Usual Care Control
Number analyzed (Participants) | 367 | 368
Participants
  Anyone smoked at home in the past 3 months | 95 | 101
  Anyone smoked in the car in the past 3 months | 117 | 125

5. Secondary Outcome: Incremental Cost Per Quit of the Intervention
Description: Establish the incremental cost per quit of the iEHR + Navigator vs. usual care arms
Time Frame: 12-months
Reporting Status: Not Posted

6. Secondary Outcome: Rates of Tobacco Use Treatment Delivery
Description: Assess the rates of tobacco treatment delivery (NRT prescription and quitline referrals) in the iEHR + Navigator arm vs. usual care, assessed by validated surveys of parents and EHR documentation
Time Frame: 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 months: Each participants adverse events were collected from the time they signed the consent to enroll in the study till they completed their follow-up data collection survey.
Arm/Group | eCEASE (iEHR + Navigator) | Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/408 | 0/409
Serious Adverse Events (participants affected / at risk) | 0/408 | 0/409
Other Adverse Events (participants affected / at risk) | 0/408 | 0/409

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04974736/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT04974736/SAP_001.pdf